CLINICAL TRIAL: NCT07364864
Title: Opioid-free Anesthesia as an Alternative to General Anesthesia in Patients Undergoing Duodenopancreatic Surgery by Laparotomy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, MD PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1072.6120.145.2025
Record Dates: First submitted 2025-12-25; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
Keywords: OFA; Opioid consumption; Opioid free anesthesia
MeSH Terms: conditions — Agnosia | interventions — Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balanced anesthesia with opioids (Active Comparator): Patients who will have duodenopancreatic surgery by laparotomy under balanced anesthesia including opioids
  Interventions: Other: Opioid
- Opioid Free Anesthesia (OFA) (Experimental): Patients who will have duodenopancreatic surgery by laparotomy under balanced anesthesia including OFA
  Interventions: Other: OFA

INTERVENTIONS:
Other: Opioid — Patients who will have duodenopancreatic surgery by laparotomy under balanced anesthesia including opioids
  Arms: Balanced anesthesia with opioids
Other: OFA — Patients who will have duodenopancreatic surgery by laparotomy under balanced anesthesia including OFA
  Arms: Opioid Free Anesthesia (OFA)

SUMMARY:
Opioid-free anesthesia is not associated with greater pain than opioid anesthesia and reduces the need for opioids in the postoperative period.

DETAILED DESCRIPTION:
Detailed Description General anesthesia using opioids is an accepted, common, and considered safe form of treatment for the patient. Opioids are associated with numerous complications, such as opioid-induced hyperalgesia (the so-called opioid paradox), and postoperative nausea, vomiting, and constipation. Modern anesthesiology, seeking alternatives to opioid-based analgesia, is increasingly turning to low-opioid and opioid-free pain management protocols. By replacing opioids with non-opioid analgesics, co-analgesics, and using regional and local anesthesia techniques, the investigators reduce or avoid the adverse effects of opioids while maintaining a satisfactory level of analgesia for the patient. Methods of administering general anesthesia without or with minimal opioid use have become particularly important in bariatric surgery, reducing the incidence of postoperative respiratory depression and excessive sedation.Opioid-free anesthesia (OFA) is a component of a multimodal, balanced general anesthesia strategy aimed at maximizing the desired analgesic effects while minimizing adverse drug reactions and side effects by utilizing the synergistic effects of various pharmacological agents in combination with regional or local anesthesia techniques. In terms of pharmacology, OFA includes opioid-free anesthesia using non-opioid analgesics - non-steroidal anti-inflammatory drugs, paracetamol, metamizole, and co-analgesics (lidocaine, magnesium, ketamine, dexmedetomidine, gabapentinoids, corticosteroids) and local anesthetics for regional anesthesia.The benefits of ketamine include improved analgesia when combined with opioids or when they are completely eliminated, a reduced incidence of chronic postoperative pain and postoperative nausea and vomiting.The additional use of lidocaine reduces pain intensity in the early postoperative period, as well as the incidence of intestinal atony, nausea and vomiting after abdominal surgery, inhibits the procedure-induced inflammatory response, and reduces the need for opioids. The group of patients to whom the OFA protocol applies includes individuals dependent on opioids, as well as patients with increased tolerance to opioids due to long-term use (pain therapy in cancer, chronic non-cancer pain). Additionally, opioids can influence the infiltration of immune cells in the tumor microenvironment and indirectly exert immunosuppressive effects, thereby participating in an additional mechanism of cancer development and escalation.Due to the increasing number of reports of cancer progression in patients undergoing surgery under general anesthesia using opioids, OFA is believed to have a favorable long-term prognostic effect, especially for oncology patients. The opioid-free protocol is also used for postoperative analgesia. It is estimated that chronic persistent postoperative pain is experienced by up to 75% of surgical patients, which has a particularly negative impact on quality of life.In our study, the investigators would like to compare the measurement of total oxycodone consumption in the postoperative period in both groups and whether the use of opioid-free anesthesia would reduce opioid consumption by 30%. The secondary objective will be to assess pain in both groups during the first 48 postoperative hours in patients undergoing pancreatic surgery who would be anesthetized with opioids and opioid-free anesthesia (patients would be randomly assigned to one group) at 1, 2, 6, 12, 24, and 48 hours after surgery. Other secondary objectives include assessing the occurrence of postoperative nausea and vomiting (PONV), adverse drug reactions, particularly cardiac arrhythmias, and the impact on persistent postoperative pain. On day 7 after surgery, each patient will receive the QOR-15 questionnaire to assess quality of life and the PQA-10 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* ASA II and III
* Patient consent to the proposed regional anesthesia
* Patient consent to participate in the study
* Surgical procedure in the pancreaticoduodenal area by laparotomy Exclusion criterion
* Patient refusal to participate in the study
* Inability to operate the PCA pump
* Lack of understanding of the NRS scale
* Hypersensitivity to anesthetics
* First- or second-degree heart block.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | up to 48 h after surgery
  oxycodone consumption in the postoperative period

SECONDARY OUTCOMES:
Pain measurment | at 1, 2, 6, 12, 24, and 48 hours after surgery
  Assessment of pain at 1, 2, 6, 12, 24, and 48 hours after surgery by NRS scale (0-10, 0 - no pain, 10 worst pain imaginable)
PONV | up to 48 h after surgery
  ponv and vomiting occurence
quality of recovery | on the 7th day after surgery
  QOR-15 questionnaire to assess quality of life and PQA-10 questionnaire. The QOR-15 is a 15 items questionnaire which provides a valid and efficient evaluation of the postoperative quality of recovery. The QoR 15 score is a score of 15 items, each scored from 0 to 10. These items assess 5 dimensions of post-operative recovery: pain, physical comfort, functional autonomy, emotions and psychological support. These 15 items represent the quality of post-operative rehabilitation in its physical and mental dimensions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Intensive Interdisciplinary Care, Collegium Medicum, Jagiellonian University, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be shared contingent upon obtaining appropriate consent from the study participants. Data will be made available only in accordance with applicable ethical and regulatory requirements.